CLINICAL TRIAL: NCT07243366
Title: Exploratory Clinical Trial of Allogeneic CD19-CAR-NK Cells in Patients With Refractory Myasthenia Gravis
Brief Title: Allogeneic CD19-CAR-NK Cells in Patients With Refractory Myasthenia Gravis
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Guangdong ProCapZoom Biosciences Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLKR-CAR-NK-I-101
Record Dates: First submitted 2025-09-09; First posted 2025-11-21 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-09

CONDITIONS: Refractory Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD19-CAR-NK Cells Group (Experimental): Allogeneic CD19-CAR-NK cells will be administered intravenously at a fixed dose, once every two weeks for a total treatment duration of 24 weeks.
  Interventions: Drug: CD19-CAR-NK Cells Injection

INTERVENTIONS:
Drug: CD19-CAR-NK Cells Injection — Allogeneic CD19-CAR-NK cells will be administered intravenously at a fixed dose, once every two weeks for a total treatment duration of 24 weeks.
  Other Names: CD19-CAR-NK Cells

SUMMARY:
This study is a single-center, prospective, nonrandom, single-arm trial.

DETAILED DESCRIPTION:
This study is a single-center, prospective, nonrandom, single-arm trial. To evaluate the clinical safety and efficacy of allogeneic CD19-CAR-NK Cells in patients with refractory myasthenia gravis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-65 years old, including the boundary value, no gender restriction;
* MGFA clinical class II-IV;
* Anti-acetylcholine-receptor antibody (AChR-Ab) shows positive;
* Willing to participate in the study, understand and sign the informed consent form (ICF).
* Baseline characteristics - all must be fulfilled:

  1. Refractory MG patients: Meet the diagnostic criteria in the Chinese Guidelines for the Diagnosis and Treatment of MG (2020 edition). On the basis of typical MG clinical features (fluctuating muscle weakness), a diagnosis can be made if any of the following three points are met, including pharmacological examination, electrophysiological characteristics, and serum anti-AChR antibody testing. Other diseases must also be excluded.
  2. Myasthenia Gravis Activities of Daily Living (MG-ADL) score ≥ 6, with ocular sub-score < 50 % of total.
* Diagnostic Criteria: Meeting any one of the following four conditions:

  1. Following an adequate dose and full course of at least two conventional immunotherapies (including both corticosteroids and non-steroidal immunosuppressants), and at least one complete treatment cycle with a biologic agent (efgartigimod, eculizumab, rituximab, or telitacicept), the post-intervention status (PIS) remains unchanged or worsens.
  2. Following an adequate dose and full course of at least two conventional immunotherapies (including both corticosteroids and non-steroidal immunosuppressants) and at least one complete treatment cycle with a biologic agent, the PIS improves, yet the MG-ADL score is still ≥6 and persists for at least six months.
  3. Following an adequate dose and full course of at least two conventional immunotherapies (including both corticosteroids and non-steroidal immunosuppressants) and at least one complete treatment cycle with a biologic agent, the PIS shows remission or improvement; however, during the regular tapering of immunotherapy drugs, the patient experiences ≥2 exacerbations per year with an MG-ADL score ≥6.
  4. Despite treatment with multiple immunotherapies-including intravenous immunoglobulin (IVIG), plasma exchange, and high-dose intravenous methylprednisolone (IVMP)-as well as aggressive infection control after a myasthenic crisis, the patient remains unable to be weaned from mechanical ventilation for more than 14 days due to respiratory muscle weakness caused by MG.
* Within 30 days before enrollment: glucocorticoids unchanged for 1 month, immunosuppressants for 3 months, pyridostigmine for 2 weeks, and stable MG-ADL score for 1 month.

Note: 1. "Two conventional immunotherapies" consist of one corticosteroid plus one non-steroidal immunosuppressant. 2. "Adequate dose for a full course" is defined as follows: 1) Corticosteroid: 0.5-1.0 mg · kg-¹ · d-¹ for ≥ 8 weeks. 2) One of the following non-steroidal immunosuppressants taken for the specified minimum duration: A. Azathioprine: 1.5-2.5 mg · kg-¹ · d-¹ in 2-3 divided doses for ≥ 24 weeks. B. Methotrexate: 15 mg once weekly for ≥ 24 weeks. C. Mycophenolate mofetil: 0.75-1.00 g twice daily for ≥ 24 weeks. D. Cyclophosphamide: 400-800 mg intravenously every week OR 100 mg/day orally in two divided doses, with a cumulative dose ≥ 15 g. E. Tacrolimus: 2-3 mg/day with at least one trough level ≥ 4.8 ng/mL for ≥ 12 weeks. F. Cyclosporine: 2-4 mg · kg-¹ · d-¹ in two divided doses, with at least one fasting trough level ≥ 100 ng/mL for ≥ 24 weeks. 3. Failure to complete the full dose and course of any one conventional immunotherapy due to contraindications, comorbidities, or inability to tolerate drug adverse effects is considered equivalent to having an inadequate response after completing a full dose and course of that conventional immunotherapy. 4. Biologic agents include efgartigimod, eculizumab, rituximab, and telitacicept.

Exclusion Criteria:

* Received IVMP, IVIG, or TPE within the 2 months before the current visit;
* Unable to cooperate in completing the MG-ADL, or QMG, or Quantitative QMG questionnaire.
* Judged by a senior clinician to have any of the following: 1)Severe or chronic urinary-tract infection; 2)History of recurrent infections; 3)Previous allergy to any human-derived biologic drug; 4)Depression, suicidal ideation, or other psychiatric disorder;
* Patients with active infection, such as herpes zoster, HIV, active tuberculosis, or active hepatitis.
* Rituximab within 6 months, eculizumab within 3 months, or efgartigimod within 1 month before enrollment.
* Receipt of any live vaccine within 3 months before screening or planned vaccination during the study.
* Subjects deemed unsuitable for participation in this trial by the investigator (e.g., severe psychiatric illness).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-11-25 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events | through study completion, an average of 1 year
  Incidence and severity of adverse events from subjects during the trial.

SECONDARY OUTCOMES:
Myasthenia Gravis Activities of Daily Living Scores | at every 2-week on-treatment visit (up to 1 month) and each follow-up (up to 1 year)
  Changes in myasthenia gravis activities of daily living scores from baseline at every 2-week on-treatment visit and each follow-up, including mean change and symptom fluctuation.
Quantitative Myasthenia Gravis Scores | at every 2-week on-treatment visit (up to 1 month) and each follow-up (up to 1 year)
  Changes in quantitative myasthenia gravis scores from baseline at every 2-week on-treatment visit and each follow-up, including mean change and symptom fluctuation.
Myasthenia Gravis Foundation of America Post-intervention Status | at every 2-week on-treatment visit (up to 1 month) and each follow-up (up to 1 year)
  Changes in myasthenia gravis foundation of America post-intervention status from baseline at every 2-week on-treatment visit and each follow-up.
AChR-antibody titers | at every 2-week on-treatment visit (up to 1 month) and each follow-up (up to 1 year)
  Changes in AChR-antibody titers from baseline at every 2-week on-treatment visit and each follow-up.
lymphocyte subsets | at every 2-week on-treatment visit (up to 1 month) and each follow-up (up to 1 year)
  Changes in lymphocyte subsets from baseline at every 2-week on-treatment visit and each follow-up.